CLINICAL TRIAL: NCT04252378
Title: Comparison of Intraoperative Opioid Consumption, Emergence Time and Hemodynamic Stability Between Ultrasound-guided Deep and Superficial Serratus Anterior Plane Block During Video-assisted Thoracoscopic Lobectomy
Brief Title: Ultrasound-guided Deep and Superficial Serratus Anterior Plane Block
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Kyungpook National University Hospital (Other)
Responsible Party: Principal Investigator, Saeyoung Kim, MD, PhD, Associate professor, Kyungpook National University Hospital
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 2019-05-003-001
Record Dates: First submitted 2020-01-31; First posted 2020-02-05 (Actual); Last update posted 2020-02-05 (Actual); Status verified 2020-02

CONDITIONS: Pain Management; Thoracotomy
MeSH Terms: conditions — Agnosia

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Deep Serratus Anterior Plane Block (Experimental): Deep Serratus Anterior Plane Block was performed just before the start of surgery after anesthetic induction through ultrasound-guidance. 20ml of 0.375% ropivacaine was slowly injected between the fascia of serratus anterior and external intercostal muscle near 5th rib.
  Interventions: Procedure: Deep Serratus Anterior Plane Block
- Superficial Serratus Anterior Plane Block (Active Comparator): Superficial Serratus Anterior Plane Block was performed just before the start of surgery after anesthetic induction through ultrasound-guidance. 20ml of 0.375% ropivacaine was slowly injected between the fascia of serratus anterior and latissimus dorsi near 5th rib.
  Interventions: Procedure: Superficial Serratus Anterior Plane Block

INTERVENTIONS:
Procedure: Deep Serratus Anterior Plane Block — Deep Serratus Anterior Plane Block was performed just before the start of surgery after anesthetic induction through ultrasound-guidance.
  Arms: Deep Serratus Anterior Plane Block
Procedure: Superficial Serratus Anterior Plane Block — Superficial Serratus Anterior Plane Block was performed just before the start of surgery after anesthetic induction through ultrasound-guidance.
  Arms: Superficial Serratus Anterior Plane Block

SUMMARY:
This study evaluates the difference of deep and superficial serratus anterior plane block on intraoperative opioid consumption, emergence time and hemodynamic stability in patients undergoing video-assisted thoracic surgery.

DETAILED DESCRIPTION:
Thoracotomy is known as one of the most painful surgery. Thus, there is a development to reduce surgical stress in terms of operation technique, which is video-assisted thoracoscopic surgery. Although it has reduced postoperative pain and complications compared with thoracotomy, VATS is still quite painful operation. Serratus plane block is a novel technique which provide analgesic effect for lateral chest wall by blocking lateral branch of intercostal nerve. Two methods were proposed to target the top and bottom of the serratus anterior muscle. However, the difference of deep and superficial serratus anterior plane block during intraoperative period has not yet been studied.

In this study, therefore, the investigators decided to assess the difference of deep and superficial serratus anterior plane block on intraoperative opioid consumption, emergence time and hemodynamic stability in patients undergoing video-assisted thoracic surgery.

ELIGIBILITY:
Inclusion Criteria:

* a) American Society of Anesthesiologists (ASA) physical status 1 or 2
* b) age 20-75 years
* c) elective three port Video-assisted thoracoscopic surgery (VATS) lobectomy.

Exclusion Criteria:

* a) a history of drug allergy for opioids or local anesthetics
* b) local infection at the injection site and systemic infection
* c) coagulopathy
* d) difficulty in understanding the study protocol
* e) refusal to participate

Ages: 20 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 56 (Estimated)
Dates: Start 2019-07-15 (Actual); Primary Completion 2020-02-29 (Estimated); Study Completion 2020-03-31 (Estimated)

PRIMARY OUTCOMES:
Intraoperative remifentanil consumption | through study completion, an average of 1 year
  Intraoperative remifentanil consumption will be checked.

SECONDARY OUTCOMES:
Emergence time | through study completion, an average of 1 year
  Emergence time is duration between the end of surgery and extubation. Emergence time will be checked.
Systolic blood pressure | through study completion, an average of 1 year
  Systolic blood pressure (mmHg) will be checked
Heart rate (HR) Heart rate | through study completion, an average of 1 year
  Heart rate (beats per minute) will be checked
Dose of rescue drugs used to control blood pressure and HR | through study completion, an average of 1 year
  Dose of rescue drugs used to control blood pressure and HR will be checked
Postoperative pain: numeric rating scale | 30 minutes later operation
  Postoperative pain will be evaluated using a numeric rating scale (0 being no pain, 10 being worst pain imaginable)

CONTACTS AND LOCATIONS:
Overall Officials: Saeyoung Kim, Principal Investigator — Kyungpook National University Hospital
Locations (1):
- Kyungpook national university hospital, Daegu, South Korea